CLINICAL TRIAL: NCT05001204
Title: 68Ga-NOTA-RM26 PET/CT for the Detection of Gastrointestinal Stromal Tumor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NMRM26
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: PET/CT; RM26; GRPR; gastrin-releasing peptide receptor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — 68Ga-NOTA-RM26

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-RM26 PET/CT (Experimental): Patients underwent whole-body PET/CT scans at 30-90 minutes after intravenous injection of 55.5-148 MBq (1.5-4 mCi) of 68Ga-NOTA-RM26.
  Interventions: Drug: 68Ga-NOTA-RM26

INTERVENTIONS:
Drug: 68Ga-NOTA-RM26 — 68Ga-NOTA-RM26 were injected into the patients before the PET/CT scans

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-RM26 in Gastrointestinal stromal tumor（GIST）patients. A single dose of 55.5 to 148 MBq(1.5-4 mCi) of 68Ga-NOTA-RM26 will be injected intravenously. Patients underwent whole-body PET/CT scans at 30-90 minutes after intravenous injection.

DETAILED DESCRIPTION:
Rm26 is a bioactive polypeptide containing 9 amino acid residues, which can specifically bind to gastrin releasing peptide receptor (GRPR, BB2 receptor). Previous studies have confirmed that there are a large number of GRPR receptors in human common types of tumors, such as lung cancer, breast cancer, prostate cancer, head and neck squamous cell carcinoma, glioma and gastrointestinal tumors. Therefore, the use of various radionuclide labeled gastrin releasing peptide receptor analogues RM26 for tumor targeted imaging and treatment greatly improves the early detection rate of tumor, and has important clinical significance and value in tumor staging, prognosis evaluation and curative effect evaluation.This prospective pilot study investigated the use of 68Ga-NOTA-RM26, an antagonist targeting gastrin-releasing peptide receptor (GRPR), for evaluating breast cancer using positron-emission tomography/computed tomography (PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients in suspicion of gastrointestinal stromal tumors by CT or ultrasonography,and being able to provide basic information and sign the written informed consent form.

Exclusion Criteria:

* The exclusion criteria included claustrophobia, pregnancy, breastfeeding, kidney or liver failure, inability to fulfill the study, and undergoing any preceding local or systemic therapies that might interfere with GRPR binding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-RM26 in gastrointestinal stromal tumor | 1 year
  The quantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (suv) of the tracer in Gastrointestinal stromal tumors will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No